CLINICAL TRIAL: NCT05927051
Title: Comparison of Different Exercise Types in Patients With Lumbal Disc Herniation
Brief Title: Effects of Exercise in Lumbal Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-20
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; McKnezie exercises; stabilization exercises
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stabilization exercises (Experimental): Core stability exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Interventions: Other: Stabilization exercises
- McKenzie exercises (Experimental): McKenzie exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Interventions: Other: McKenzie exercises
- Home exercises (Experimental): Home exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Interventions: Other: Home exercises

INTERVENTIONS:
Other: Stabilization exercises — Core stability exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Arms: Stabilization exercises
Other: McKenzie exercises — McKenzie exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Arms: McKenzie exercises
Other: Home exercises — Home exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks
  Arms: Home exercises

SUMMARY:
Lumbar disc herniation, which causes 5% of all low back pain, is the rupture of the annulus fibrosis in the intervertebral disc in the lumbar region and the protrusion of the nucleus pulposus at various degrees, and as a result, the spinal cord or the nerves arising from it are compressed.Aerobic exercise is one of the most important elements in low back pain rehabilitation.Many studies have shown that individuals with low back pain have low muscle strength of the back extensors and flexors when compared to individuals who do not show symptoms, and that these muscles are strong and their aerobic fitness is high, minimizing trauma-related musculoskeletal damage.The aim of this study is to examine the effect of core stabilization exercises on functionality and core muscles in patients with LDH.

DETAILED DESCRIPTION:
n general, low back pain is defined as pain that negatively affects comfort in the lower back and/or legs. Low back pain lasting less than 6 weeks is defined as acute, 6-12 weeks as subacute, and lasting longer than 12 weeks as chronic low back pain. Depending on the low back pain of the people, the activity level decreases and therefore aerobic fitness is negatively affected. As a result of this negative impact, chronic conditions pose a risk in terms of cardiovascular disease and lead to a decrease in work capacity. Therefore, aerobic exercise is one of the most important elements in low back pain rehabilitation. In our country, training on regular exercise habits and waist protection methods is very low. Most patients do not apply to health institutions unless symptoms become severe.Many studies have shown that individuals with low back pain have low muscle strength of the back extensors and flexors when compared to individuals who do not show symptoms, and that these muscles are strong and their aerobic fitness is high, minimizing trauma-related musculoskeletal damage.

Core stabilization and strengthening has been the subject of research in the 1980s. The purpose of these exercises is to increase trunk stability and aerobic capacity. It is used to find and maintain the neutral position, to reduce ligament, tendon and joint tension, to reduce the load on discs and facet joints, to increase functional stability in low back pain, disc herniation and post-operative rehabilitation of patients.The researchers' studies have shown that ultrasound imaging is reliable in measuring TrA thickness in both healthy subjects and low back patients.

The aim of this study is to examine the effect of core stabilization exercises on functionality and core muscles in patients with LDH.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 to 65
* Patients who have diagnosed with LDH

Exclusion Criteria:

* Patients who were pregnant
* diagnosed with malignancy
* had changes of medical treatment in the last 3 months
* had dysfunction that limited physical activity such as severe neurological impairment,
* immobility or cooperation deficits
* had regular exercise habit (minimally three days in a week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Core muscle thickness | 2 minutes
  Ultrasonographic images of the transversus abdominis (TrA), lumbar multifidus (MF) and Gluteus maximus (G max) muscles will be acquired using B mode (TOSHIBA Aplio 300, Japan).

SECONDARY OUTCOMES:
Visual Analog Scale | 1 minute
  Pain Severity; It will be evaluated with a 10 cm Visual Analogue Scale (VAS). Patients are told what the numbers on the horizontal line mean, 0 is no pain, 10 is the most severe pain in life, and 5 is moderate pain, and they are asked to describe the severity of their pain on the scale.
Modified Oswerty Inquiry | 2 minutes
  Functional Disability Measurement; The evaluation will be made using the Turkish version of the Modified Oswestry Inquiry Form. Turkish validity and reliability were determined by Edibe Yakut et al. (2004) by In the evaluation of the Oswestry scale, scoring for each question is A=0 B=1 C=2 D=3 E=4 F=5 points. Questions that the patient does not answer will not be evaluated. Evaluation is made on the basis of the questions answered. Patient score =(Patient score/Maximum possible score)*100

CONTACTS AND LOCATIONS:
Locations (1):
- Songül Bağlan Yentür, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Optimizing performance by improving core stability and core strength — http://pubmed.ncbi.nlm.nih.gov/19026017/
- See also: Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care — http://pubmed.ncbi.nlm.nih.gov/16550447/